CLINICAL TRIAL: NCT03246568
Title: Renal Artery Sympathetic Denervation by Catheter Ablation After Pulmonary Vein Isolation for Persistent Atrial Fibrillation
Brief Title: Renal Nerve Denervation After Pulmonary Vein Isolation for Persistent Atrial Fibrillation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: no funding to purchase study device
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Bryan Ping Yen YAN, Associate Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CUHK-CARD-2017-RND
Record Dates: First submitted 2017-08-09; First posted 2017-08-11 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Atrial Fibrillation
Keywords: Ablation; Renal Denervation; Cryoballoon
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Research on the Basis of Earlier Theory Renal artery sympathetic denervation (RND) by catheter ablation has been shown in a preliminary study to improve outcome of electrical isolation of the pulmonary vein (PVI) in patients with paroxysmal and/or persistent AF with concomitant refractory hypertension and the same group later showed renal sympathetic denervation improved outcome of PVI in the cohort of paroxysmal and/or persistent AF patients with moderate hypertension. In patients with renal impairment, RND also conferred benefit in reducing AF recurrence after PVI.The initial indication for catheter-based RND is for blood pressure control in patients with resistant hypertension. Early data from clinical trials without sham controls was promising - demonstrating large blood pressure reductions in patients with treatment-resistant hypertension.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulmonary vein isolation alone (Active Comparator): PVI by cryo-balloon ablation without linear ablation
  Interventions: Procedure: Pulmonary vein isolation
- Renal nerve denervation (Experimental): PVI by cryo-balloon ablation without linear ablation plus bilateral RND using a multi-electrode renal denervation catheter.
  Interventions: Procedure: Renal Nerve Denervation; Procedure: Pulmonary vein isolation

INTERVENTIONS:
Procedure: Renal Nerve Denervation — Bilateral renal denervation using a multi-polar radiofrequency ablation catheter (Symplicity™ Spyral Cather, Medtronic) in the right and left main, branch, and accessory renal arteries in vessels ranging in diameter between 3 and 8 mm.
  Other Names: Renal artery sympathetic nerve denervation; RND
  Arms: Renal nerve denervation
Procedure: Pulmonary vein isolation — PVI by cryo-balloon ablation without linear ablation
  Other Names: PVI

SUMMARY:
Atrial fibrillation (AF) is the most common arrhythmia and it is associated with significant morbidity and mortality. Electrical isolation of the pulmonary vein (PVI) by radiofrequency energy or cryoablation has been shown to be an effective treatment of AF by reducing morbidity, improving quality of life and functional capacity.

Renal artery sympathetic denervation (RND) by catheter ablation has been shown in a preliminary study to improve outcome of PVI in patients with paroxysmal and/or persistent AF with concomitant refractory or moderate hypertension. In patients with renal impairment, RND also conferred benefit in reducing AF recurrence after PVI. The initial indication for catheter-based RND is for blood pressure control in patients with resistant hypertension. However, a recent study failed to show significant difference in blood pressure reduction by RND. Therefore, the effect of RND on AF suppression may be independent of blood pressure control. Possible mechanisms of RND on AF may include risk factors modification and anti-arrhythmic effect.

DETAILED DESCRIPTION:
This prospective randomized study aimed to evaluate the effect of RDN added to PVI for persistent AF. Study will be performed in accordance with Declaration of Helsinki.

Study Hypothesis: Catheter based RDN can prevent recurrence of AF in patient with persistent AF undergoing PVI by mechanism not related to hypertension control.

Primary outcome measure: Freedom from documented AF episodes post PVI as defined by longer than 30 seconds of AF recorded by implantable loop recorder 2 to 18 months after procedure with or without antiarrhythmic medication.

Sample Size:

This is an exploratory study, the sample size calculation will not be applied and arbitrary assign 20 subjects to each arm will be adopted.

Randomization Arms:

Patients are randomized in 1:1 fraction to one of the following arms:

1. PVI by cryo-balloon ablation without linear ablation;
2. PVI by cryo-balloon ablation without linear ablation plus bilateral RND using a multi-electrode renal denervation catheter.

ELIGIBILITY:
Inclusion Criteria:

1. Patients age is 18 years or greater;
2. Patients undergoing a first-time ablation procedure for AF;
3. Patients with persistent AF;
4. Persistent AF will be defined as a sustained episode lasting > 7 days and less than 3 years.
5. Patients with symptomatic AF that is refractory to at least one antiarrhythmic medication;
6. Symptomatic patients are those who have been aware of their AF at any time within the last 5 years prior to enrollment. Symptoms may include, but are not restricted to, palpitations, shortness of breath, chest pain, fatigue, left ventricular dysfunction, or other symptoms, or any combination of the above.
7. At least one episode of persistent AF must have been documented by ECG, Holter, loop recorder, telemetry, trans telephonic monitoring (TTM), or implantable device within last 2 years of enrollment in this investigation.

Exclusion Criteria:

1. Patients with paroxysmal AF;
2. Paroxysmal AF will be defined as a sustained episode lasting < 7 days.
3. Patients with long-standing persistent AF;
4. Long-standing persistent AF will be defined as a sustained episode lasting more than 3 years;
5. Patients for whom cardioversion or sinus rhythm will never be attempted/pursued;
6. Patients with AF felt to be secondary to an obvious reversible cause;
7. Patients with contraindications to systemic anticoagulation with heparin or warfarin or a direct thrombin inhibitor;
8. Patients with left atrial size ≥ 60 mm (2D echocardiography, parasternal long axis view);
9. Patients with more than 50% renal artery stenosis identified by duplex ultrasound or renal angiogram;
10. Patients in whom a renal stent has been in place for less than3 months;
11. Patients with prior renal artery stent placement, the artery segment beyond the stent margins must be able to accommodate treatments;
12. Patients with the treatment zone for denervation in the renal artery have areas of atheroma, severe fibromuscular dysplasia, calcification, and aneurysm that cannot be avoided;
13. Patients with renal dysfunction as demonstrated by an estimated glomerular filtration rate less than 45 mL/min per 1.73 m2 are excluded from both studies;
14. Pregnant women;
15. Participation in another interventional study;
16. Patient with contraindication to left ventricle catheterization by a retrograde aortic approach (eg mechanical aortic valve, severe aortic stenosis and aortic dissection).
17. Patient with systolic blood pressure <100mmHg.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-09-17 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Freedom from documented AF episodes post PVI by implantable loop recorder by implantable loop recorder. | 2 to 18 months after procedure
  Freedom from documented AF episodes post PVI as defined by longer than 30 seconds of AF recorded by implantable loop recorder 2 to 18 months after procedure with or without antiarrhythmic medication.

SECONDARY OUTCOMES:
Freedom from documented atrial arrhythmia episodes post PVI by implantable loop recorder. | 2 to 18 months after procedure
  Freedom from documented atrial arrhythmia episodes post PVI as defined by longer than 30 seconds of atrial arrhythmia recorded by implantable loop recorder 2 to 18 months after procedure with or without antiarrhythmic medication.
Freedom from symptomatic AF episodes post PVI by implantable loop recorder. | 2 to 18 months after procedure
  Freedom from symptomatic AF episodes post PVI as defined by longer than 30 seconds of AF recorded by implantable loop recorder 2 to 18 months after procedure with or without antiarrhythmic medication.
Freedom from symptomatic atrial arrhythmia episodes post PVI by implantable loop recorder. | 2 to 18 months after procedure
  Freedom from symptomatic atrial arrhythmia episodes post PVI as defined by longer than 30 seconds of atrial arrhythmia recorded by implantable loop recorder 2 to 18 months after procedure with or without antiarrhythmic medication.
Freedom from documented AF episodes post PVI by hand-held smartphone device. | 2 to 18 months after procedure
  Freedom from documented AF episodes post PVI as defined by 30 seconds of AF recorded by hand-held smartphone device (i.e. Cardiio Rhythm iPhone AF-detection system or AliveCor single-lead ECG device) 2 to 18 months after procedure with or without antiarrhythmic medication.
The mean blood pressure as measured by 24-hour ambulatory blood pressure monitoring. | 18 months
  The mean blood pressure as measured by 24-hour ambulatory blood pressure before and after ablation up to 36 months.
Incidence of peri-procedural complications. | 18 months
  Incidence of peri-procedural complications, including stroke, PV stenosis, cardiac perforation, phrenic nerve palsy, esophageal injury and death.
Procedure duration | duing procedure
  Procedure duration
Fluoroscopy time during procedure | dueing procedure
  Fluoroscopy time during procedure
Number of repeat procedures | 18 months
  Number of repeat procedures

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Ping Yen YAN, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No